CLINICAL TRIAL: NCT02486094
Title: Study Of PRoliferation and Apoptosis in Rectal caNcer as Predictive and Prognostic biOmarkers: a Histopathology and Imaging Analysis
Brief Title: Study of PRoliferation and Apoptosis in Rectal Cancer, Predictive & Prognostic biOmarkers: Histopathology and Imaging
Acronym: SOPRANO
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: The Royal College of Surgeons of England (Other); Croydon Health Services NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 4324
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2015-06

CONDITIONS: Neoplasms; Colorectal Neoplasms; Rectal Diseases; Gastrointestinal Neoplasms
Keywords: Imaging, Magnetic Resonance; Rectal Cancer; Apoptosis; Proliferation; Cancer; Tissue Study
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Rectal Diseases; Gastrointestinal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pre-treatment biopsy and post surgical tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
This study tests biopsy and tissue from patients who have been treated for primary rectal cancer at the Royal Marsden Hospital between 2011 and 2013, who have an mrTRG score at post-chemoradiotherapy MRI. It is a retrospective pilot study to determine the apoptotic and proliferative index count pre and post chemoradiotherapy.

DETAILED DESCRIPTION:
The investigators hope to validate the apoptotic and proliferative index as a predictive response marker and lend support to mrTRG as a putative prognostic tool in the treatment pathway for rectal cancer patients. Even though this is a retrospective study, the investigators hope that pre-treatment apoptotic and proliferative scores will correlate to post treatment response and mrTRG scores. In doing so, the investigators can predict how patients will respond to treatment from initial diagnostic biopsies and foresee a patients individual treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with primary adenocarcinoma of the rectum (diagnosed on tissue biopsy and disease spread assessed on CT and MRI).
* Tumours must be considered sufficiently high-risk to require pre-operative chemoradiotherapy followed by surgery.
* Patients must have had a pre- and post-treatment MRI scan of the rectum and pelvis.
* We must have access to stored tissue for each patient

Exclusion Criteria:

* No pre-operative radiotherapy
* Patients with synchronous tumours
* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer, diagnosed between 2011 and 2013, who have had an mrTRG score in a post-radiotherapy MRI scan.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09-01 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Apoptotic index, Ki67 and Geminin in cells per mm cubed from diognostic biopsy | Tissue removed at diagnosis (approximately 15 weeks prior to surgery)
  Tissue biopsy taken at endoscopy to confirm cancer diagnosis is studied
Apoptotic index, Ki67 and Geminin in cells per mm cubed from resected tumour | Tissue removed during operation
  Tissue removed during surgery (to resect tumour) is studied

SECONDARY OUTCOMES:
Time to local recurrence | At one and three years
Disease Free Survival (DFS) | At one and three years
Overall Survival (OS) | At one and three years

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey, United Kingdom